CLINICAL TRIAL: NCT05108961
Title: Randomized Propective Study Evaluating the Impact of an Acupuncture Session in Healthy Volunteers on the Kinetics of Cerebral Activity Using the Bispectral Index (BIS)
Brief Title: Evaluation of the Impact of an Acupuncture Session in Healthy Volunteers on the Kinetics of Cerebral Activity Using the Bispectral Index (BIS)
Acronym: Bisprectral2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Collaborators: European Clinical Trial Experts Network (Other); Clinique saint martin Pessac (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021-A01814-37
Record Dates: First submitted 2021-10-15; First posted 2021-11-05 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Acupuncture; Healthy Volunteers
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture arm (Experimental): One session of acupuncture with precise acupuncture points
  Interventions: Procedure: Acupuncture; Behavioral: A digital stress scale; Behavioral: a relaxation questionnaire; Diagnostic Test: Bispectral Index
- Sham acupuncture arm (Sham Comparator): One session of sham acupunture (needles inserted 1 mm, outside the acupuncture points)
  Interventions: Behavioral: A digital stress scale; Behavioral: a relaxation questionnaire; Diagnostic Test: Bispectral Index
- Control arm (Placebo Comparator): One session where no needles are inserted, the subject lies down under the same conditions as group 1 and 2
  Interventions: Behavioral: A digital stress scale; Behavioral: a relaxation questionnaire; Diagnostic Test: Bispectral Index

INTERVENTIONS:
Procedure: Acupuncture — one session with precise acupunture points
  Arms: Acupuncture arm
Behavioral: A digital stress scale — The digital stress scale before and after the session: Oral digital scale. The doctor asks the participant to quantify their anxiety on a virtual scale ranging from 0 (absent anxiety) to 10 (maximum anxiety imaginable)
Behavioral: a relaxation questionnaire — The Global Relaxation Questionnaire after the session: Dovero Global Relaxation Scale
Diagnostic Test: Bispectral Index — BIS is based on an EEG analysis algorithm

SUMMARY:
To be able to have data on brain activity during an acupuncture session, this pilot study is necessary to evaluate the kinetics of the bispectral index. This research aims to evaluate the kinetics of the bispectral index in healthy volunteers during an acupuncture session, Sham acupuncture or resting in a lying position.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Over 18 years old and less than 65.
* Having given his express consent
* Affiliated to a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Medical history of psychiatric disorders
* Psychotropic treatment
* narcolepsy
* Obstructive sleep apnea syndrome
* Symptoms that may correspond to COVID 19
* Nickel allergy
* Refusal to participate in the study
* Protected subjects : Adults under guardianship, curatorship or other legal protection deprived of their liberty by judicial or administrative decision
* Pregnant, breastfeeding or parturient woman
* Subject hospitalized without consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Bispectral Index | 35 minutes
  Bispectral Index (BIS) measured every second for 35 min through an EEG

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Saint Martin, Pessac, France